CLINICAL TRIAL: NCT04151121
Title: Mindfulness Based Intervention in Patients With Persistent Pain in Chest (MIPIC) of Non-Cardiac Cause - a Feasibility Randomised Control Study
Brief Title: Mindfulness in Chest Pain - a Feasibility Randomized Controlled Study
Acronym: MIPIC
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Royal Brompton & Harefield NHS Foundation Trust (Other)
Collaborators: University of Oxford (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 253106
Record Dates: First submitted 2019-10-30; First posted 2019-11-05 (Actual); Last update posted 2022-05-02 (Actual); Status verified 2022-04

CONDITIONS: Chest Pain
Keywords: chest pain; non-cardiac; mindfulness
MeSH Terms: conditions — Chest Pain | interventions — Mindfulness-Based Cognitive Therapy

STUDY DESIGN:
Intervention Model Description: Simple 1:1 randomization.
Who Masked: Outcomes Assessor
Masking Description: The research staff conducting the outcome follow-up will be blinded to the randomization.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention (Experimental): The participants will receive MBCT (Mindfulness-Based Cognitive Therapy) as 2-hourly sessions over 8-weeks including a 6-hour session at the end of 6th week. The MBCT will be adapted for chest pain.
  Interventions: Behavioral: MBCT (Mindfulness Based Cognitive Therapy)
- Control group (No Intervention): These participants will continue to receive any treatment (or no treatment) by their primary care physicians.

INTERVENTIONS:
Behavioral: MBCT (Mindfulness Based Cognitive Therapy) — MBCT is recognized behavior therapy for patients with recurrent depression. The program will be adapted for patients with chest pain.
  Arms: Intervention

SUMMARY:
Non-cardiac chest pain (NCCP) is a common symptom in clinical practice with no satisfactory treatment. We plan to perform a feasibility randomized controlled trial (RCT) to explore the role of mindfulness therapy in patients with NCCP to ascertain the number of patients who would be willing to enroll and complete the mindfulness intervention. This will allow us to develop and refine the adaption of mindfulness therapy as well as assess the compliance.

DETAILED DESCRIPTION:
Chest pain is a common condition in primary care with the lifetime prevalence of no cardiac cause (NCCP) being 20-33 percent compared to 6-7 percent for cardiac chest pain. The latter patients obtain appropriate medical and interventional treatment but those with NCCP are often left with persistent symptoms, psychological distress, impaired quality of life, high unemployment, work absenteeism, and high use of healthcare resources. They are often treated with analgesics, proton-pump inhibitors, anxiolytics, but generally with little benefit.

Mindfulness has grown in popularity in the last 2-3 decades as an accepted form of behavior therapy for the treatment of stress and depression. Several RCTs have been performed in patients with chronic pain, but none specific to chest pain. They have been heterogeneous in nature with low-quality evidence for improvement of pain with mindfulness. There is thus a requirement for larger, well-designed and rigorous RCTs in patients with chronic pain, including those with NCCP.

With this feasibility RCT study, the investigators would like to obtain more information about some uncertainties that would allow them to conduct a larger, well-designed RCT. The investigators plan to recruit 50 participants from all those who have attended the chest pain clinic in the previous 12-months and randomize them in a simple 1:1 manner into receiving Mindfulness-based Cognitive Therapy (MBCT) therapy (intervention arm) or usual treatment by their general practitioner (control arm). The participants will undergo a basic clinical assessment with symptoms, heart-rate, blood pressure, height, body weight, cardiovascular risk factors. They will be required to complete different questionnaires to assess their chest pain limitation and frequency, general and cardiac-specific anxiety, mindfulness, quality of life, and health-related resource utilization at baseline and after completion of MBCT or usual treatment.

ELIGIBILITY:
Inclusion Criteria:

* Attendance to the chest pain clinic within the last 12 months and no cardiac cause for chest pain were identified.
* Have persistent chest pain symptoms on or after usual treatment
* Ability to carry out the 8-week mindfulness course and required home practice.
* Able to understand verbal and written English.

Exclusion Criteria:

* Acute presentation with ECG changes and/ or raised enzymes at any time prior to enrolment.
* Known history of coronary artery disease.
* Under active psychiatric care or waiting for a psychological assessment or have received a prescription of a new psychoactive drug within the previous 3 months.
* Undergoing any other form of counselling or behaviour therapy.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 32 (Actual)
Dates: Start 2019-12-01 (Actual); Primary Completion 2020-09-30 (Actual); Study Completion 2021-03-30 (Actual)

PRIMARY OUTCOMES:
Willingness to participate in mindfulness-based behaviour therapy | 8 months
  To assess the number of patients with persistent chest pain without a heart condition who would be willing (and consent) to participate in mindfulness-based behaviour therapy
Compliance with mindfulness-based behavior therapy | 8 months
  To assess compliance with the mindfulness program by participation in the 8-week sessions and home practice. Each participant will be given a worksheet to complete for home practice and their experience.

SECONDARY OUTCOMES:
Persistent chest pain | 8-months
  To assess the number of patients diagnosed as non-cardiac chest pain who have persistent chest pain. This will be ascertained during the initial phone call by the research team. It will be further assessed in terms of physical limitation and frequency by the Seattle Angina Questionnaire at baseline and at follow-up. However, as this is a feasibility study, it is not powered to demonstrate statistically significant changes.
Prevalence of general anxiety and depression | 8- months
  To assess the prevalence of general anxiety and depression by means of Hospital Anxiety and Depression Scale questionnaire at baseline and at follow-up. However, as this is a feasibility study, it is not powered to demonstrate statistically significant changes.
Prevalence of cardiac anxiety | 8 months
  To assess the prevalence of heart-focussed anxiety with Cardiac Anxiety Questionnaire (CAQ) at baseline and follow-up. However, as this is a feasibility study, it is not powered to demonstrate statistically significant changes.
State of mindfulness | 8-months
  Each participant's state of mindfulness will be assessed using Five Facet Mindfulness Questionnaire at baseline and follow-up. However, as this is a feasibility study, it is not powered to demonstrate statistically significant changes.
Generic health related quality of life | 8-months
  Each participant's quality of life, including limitations in bodily and mental functioning associated with persistent chest pain, will be assessed by means of EuroQuol-5 questionnaire. However, as this is a feasibility study, it is not powered to demonstrate statistically significant changes.
Health resource utilization | 8-months
  The study will evaluate the utilization of health resources in terms of the number of visits to the hospital (as in-patient or out-patient) and primary care using Adult Service Use Schedule (AD-SUS) at baseline and follow-up.

CONTACTS AND LOCATIONS:
Overall Officials: Tarun K Mittal, MD, FRCR, Principal Investigator — Royal Brompton & Harefield NHS Foundation Trust
Locations (1):
- Harefield Hospital, London, Middlesex, United Kingdom

IPD SHARING:
Plan to Share IPD: Yes
We plan to share individual participant data with any other researcher that underlie results in a publication.
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: Data will be available after study publication for a period of 3 years.
Access Criteria: Data access requests will be reviewed by the study investigators. Requestors will be required to sign a Data Access Agreement.

REFERENCES:
- [Background] Hoorweg BB, Willemsen RT, Cleef LE, Boogaerts T, Buntinx F, Glatz JF, Dinant GJ. Frequency of chest pain in primary care, diagnostic tests performed and final diagnoses. Heart. 2017 Nov;103(21):1727-1732. doi: 10.1136/heartjnl-2016-310905. Epub 2017 Jun 20. PMID 28634285
- [Background] Tyrer P, Tyrer H, Morriss R, Crawford M, Cooper S, Yang M, Guo B, Mulder RT, Kemp S, Barrett B. Clinical and cost-effectiveness of adapted cognitive behaviour therapy for non-cardiac chest pain: a multicentre, randomised controlled trial. Open Heart. 2017 May 16;4(1):e000582. doi: 10.1136/openhrt-2016-000582. eCollection 2017. PMID 28674627
- [Background] Mittal TK, Pottle A, Nicol E, Barbir M, Ariff B, Mirsadraee S, Dubowitz M, Gorog DA, Clifford P, Firoozan S, Smith R, Dubrey S, Chana H, Shah J, Stephens N, Travill C, Kelion A, Pakkal M, Timmis A. Prevalence of obstructive coronary artery disease and prognosis in patients with stable symptoms and a zero-coronary calcium score. Eur Heart J Cardiovasc Imaging. 2017 May 1;18(8):922-929. doi: 10.1093/ehjci/jex037. PMID 28379388
- [Background] Kuyken W, Warren FC, Taylor RS, Whalley B, Crane C, Bondolfi G, Hayes R, Huijbers M, Ma H, Schweizer S, Segal Z, Speckens A, Teasdale JD, Van Heeringen K, Williams M, Byford S, Byng R, Dalgleish T. Efficacy of Mindfulness-Based Cognitive Therapy in Prevention of Depressive Relapse: An Individual Patient Data Meta-analysis From Randomized Trials. JAMA Psychiatry. 2016 Jun 1;73(6):565-74. doi: 10.1001/jamapsychiatry.2016.0076. PMID 27119968
- [Background] Chambers JB, Marks EM, Hunter MS. The head says yes but the heart says no: what is non-cardiac chest pain and how is it managed? Heart. 2015 Aug;101(15):1240-9. doi: 10.1136/heartjnl-2014-306277. Epub 2015 Apr 16. No abstract available. PMID 25882503
- [Background] Kisely SR, Campbell LA, Yelland MJ, Paydar A. Psychological interventions for symptomatic management of non-specific chest pain in patients with normal coronary anatomy. Cochrane Database Syst Rev. 2015 Jun 30;2015(6):CD004101. doi: 10.1002/14651858.CD004101.pub5. PMID 26123045
- [Background] Ludwig DS, Kabat-Zinn J. Mindfulness in medicine. JAMA. 2008 Sep 17;300(11):1350-2. doi: 10.1001/jama.300.11.1350. No abstract available. PMID 18799450
- [Background] Robertson N, Javed N, Samani NJ, Khunti K. Psychological morbidity and illness appraisals of patients with cardiac and non-cardiac chest pain attending a rapid access chest pain clinic: a longitudinal cohort study. Heart. 2008 Mar;94(3):e12. doi: 10.1136/hrt.2006.100537. Epub 2007 May 31. PMID 17540685
- [Background] Kabat-Zinn J. An outpatient program in behavioral medicine for chronic pain patients based on the practice of mindfulness meditation: theoretical considerations and preliminary results. Gen Hosp Psychiatry. 1982 Apr;4(1):33-47. doi: 10.1016/0163-8343(82)90026-3. PMID 7042457
- [Derived] Mittal TK, Evans E, Pottle A, Lambropoulos C, Morris C, Surawy C, Chuter A, Cox F, de Silva R, Mason M, Banya W, Thakrar D, Tyrer P. Mindfulness-based intervention in patients with persistent pain in chest (MIPIC) of non-cardiac cause: a feasibility randomised control study. Open Heart. 2022 May;9(1):e001970. doi: 10.1136/openhrt-2022-001970. PMID 35545356